CLINICAL TRIAL: NCT02275819
Title: Exercise Training in Heart Failure: Structural and Functional Cardiac Remodeling
Brief Title: Exercise Training in Heart Failure: Changes in Cardiac Structure and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1423-P
Record Dates: First submitted 2014-10-03; First posted 2014-10-27 (Estimated); Results first posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure
Keywords: Heart Failure; Exercise; Echocardiography
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Non-randomized case control study with two groups. One group received exercise and the controls did not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): Will not receive intervention with exercise
- Intervention group (Active Comparator): 2 groups will receive 2 different types of therapy (exercise or Inspiratory Muscle Therapy)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise (walking 3 times a week for 60 minutes) or Inspiratory Muscle Therapy (breathing against an inspiratory resistive load 3 times a week for up to 60 minutes)
  Arms: Intervention group

SUMMARY:
This is a research study being conducted to better understand the impact of exercise training on changes on the structure and function of the heart. Exercise training in patients with heart failure has been shown to be beneficial at decreasing symptoms of heart failure and improving overall functional capacity or capacity to exercise. However the mechanisms responsible for this are still unclear. This study will look specifically at how exercise creates changes within the hearts filling ability, the hearts pumping strength as well as the hearts ability to rebuild.

DETAILED DESCRIPTION:
Prevalence of systolic heart failure (HF) is high among the growing population of older adults. Progressive cardiac remodeling and deteriorating cardiac output have been implicated as key factors underlying HF-related exercise intolerance and quality of life. Even after implementing medical and device therapies that moderate remodeling, exercise tolerance remains impaired. While exercise training has been demonstrated to improve exercise capacity, mechanisms facilitating this benefit remain unclear. Peripheral adaptations in the skeletal muscle and vasculature provide at least some benefit, however reverse cardiac remodeling (beyond effects of pharmacological and device therapies) may be additive. The investigators propose to study the impact of 2 different types of exercise on cardiac morphology as well as systolic and diastolic performance and related functional gains. The investigators will compare traditional aerobic training to a novel regimen of inspiratory muscle training (IMT). IMT is a specific type of exercise training that may be particularly useful for frail, infirmed HF patients who are unlikely to tolerate aerobic training. Effects of IMT on remodeling have not been previously studied.

The proposed echocardiography pilot study builds on a funded VA Merit F0834-R "Exercise Therapy to Reduce Heart Failure Symptoms; Sorting Mechanisms of Benefit" (Exercise therapy) PI, Forman that compares different modes of exercise training in older (age 50yrs) systolic (EF 45%) HF patients. The original study assesses peripheral mechanisms affected by exercise training, but was not designed to assess cardiac remodeling. The proposed pilot study provides a vital complementary analysis, i.e., it adds assessments of cardiac remodeling as well as related changes in systolic and diastolic performance.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) class II or III for the previous three months despite a minimum of 6 weeks of optimal treatment.
* Age >50 years.
* Left Ventricular Ejection Fraction (LVEF)<45% (by echocardiogram or radionucleotide imaging study within 6 months of enrollment). If a patient has initiated or received any therapy that might improve the ejection fraction, the qualifying EF must be assessed after the patient is on a stable dose of these therapies. Additionally the LVEF of <45% will be confirmed with a brief echocardiogram prior to randomization. If LVEF is not 45%, the patient will not be enrolled in to the study.
* Optimal therapy according to the American Heart Association (AHA)/American College of Cardiology (ACC) and the Heart Failure Society of America (HFSA) Heart Failure (HF) guidelines, including treatment with an angiotensin-converting-enzyme (ACE) Inhibitor (or an angiotensin receptor blocker) and beta-blocker therapy (for at least 6 weeks), or have documented reason for variation, including medication intolerance, contraindication, patient preference, or personal physician's judgment.

In addition to the above we have now added patients with heart failure with preserved ejection fraction (similar to the parent study )pending Institutional Review Board (IRB) review.

Exclusion Criteria:

* Major cardiovascular event or procedure within the prior 6 weeks.
* Dementia.
* Severe chronic obstructive pulmonary disease (COPD) (FEV1<50%), peripheral vascular disease (PVD), and/or Anemia.
* End-stage malignancy.
* Severe valvular heart disease.
* Orthopedic exercise limitation.
* Women who are pregnant, breastfeeding, or likely to become pregnant within the next 6 months.
* Psychiatric hospitalization within the last 3 months.
* Implantable Cardioverter Defibrillator (ICD) device with heart rate limits that prohibit exercise assessments or exercise training. Referring physicians will be provided with an opportunity to reprogram devices so that patients can participate.
* Chronic ethyl alcohol (ETOH) or drug dependency.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Aragam, MD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at VA Boston Healthcare System cardiology related clinics from 6/6/2016 to 12/21/2018. As per the protocol the recruitment was supposed to begin in 2014. Unfortunately there were a number of issues including the fact that the parent study moved to Pittsburgh and we were not able to start recruitment till 2016.
Pre-assignment Details: 13 participants were consented but only 11 were enrolled. Two were excluded from randomization due to subsequent echocardiogram or pulmonary function screening not meeting enrollment criteria. One was withdrawn after enrollment due to increasing symptoms of heart failure.
  Due to the small number of participants enrolled in each of the active intervention arms we combined participants from both intervention groups and analyzed against the controls.
Groups:
- Intervention Group: 2 groups will receive 2 different types of exercise
Period: Overall Study
Arm/Group | Control | Intervention Group
Started | 5 | 6
Completed | 5 | 5
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention Group | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (8.4) | 67.2 (4.4) | 68.4 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular Systolic Function.
Description: Change in left ventricular ejection fraction.
Time Frame: Baseline and endpoint at 3-5 months
Measure: Mean (Standard Deviation); unit: percent LVEF
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 5 | 5
percent LVEF | .82 (3.54) | -1.90 (1.14)
Statistical Analysis 1: Comparison: Control vs Intervention Group; Test type: Superiority; p = .14, t-test, 2 sided

2. Primary Outcome: Change in Left Ventricular Structure.
Description: Change in left ventricular mass.
Time Frame: Baseline and endpoint at 3-5 months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 5 | 5
grams | -34.8 (49.8) | 3.1 (40.8)
Statistical Analysis 1: Comparison: Control vs Intervention Group; Test type: Superiority; p = .22, t-test, 2 sided

3. Primary Outcome: Change in Diastolic Function.
Description: Change in mitral annular early diastolic velocity (e')
Time Frame: Baseline and endpoint at 3-5 months
Measure: Mean (Standard Deviation); unit: centimeters/second
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 5 | 5
centimeters/second | .31 (.68) | -1.07 (1.42)
Statistical Analysis 1: Comparison: Control vs Intervention Group; Test type: Superiority; p = .12, t-test, 2 sided

4. Primary Outcome: Change in Left Ventricular (LV) Diastolic Function
Description: Change in the ratio of early mitral in-flow velocity (E) to mitral annular early diastolic velocity (e')
Time Frame: Baseline and endpoint at 3-5 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 5 | 5
ratio | -1.85 (3.06) | 2.68 (3.49)
Statistical Analysis 1: Comparison: Control vs Intervention Group; Test type: Superiority; p = .08, t-test, 2 sided

5. Primary Outcome: Change in Right Ventricular Function
Description: Change in tricuspid annular tissue doppler velocity
Time Frame: Baseline and endpoint at 3-5 months
Measure: Mean (Standard Deviation); unit: centimeters/second
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 5 | 5
centimeters/second | 0.16 (1.04) | -0.70 (2.05)
Statistical Analysis 1: Comparison: Control vs Intervention Group; Test type: Superiority; p = 0.43, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected while participants were enrolled from enrollment until collection of the final study endpoint at 3-5 months.
Arm/Group | Control | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 4/5
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=5) | Intervention Group (N=5)
ER Visit (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient had flu like symptoms and started coughing up blood. Patient treated with Tamiflu and sent home.
HF exacerbation (Cardiac disorders) | 0 (0) | 1 (1) — Patient reported swelling and edema in legs. Reported to ER and was admitted.
Low BP (Cardiac disorders) | 0 (0) | 1 (1) — Patient had low BP of 70/50 during a study visit. All other measures were in normal range. Had been taking additional diuretic and additional exercise. Patient was evaluated by cardiologist and sent home for dehydration.
A-fib Hospitalization (Cardiac disorders) | 0 (0) | 1 (1) — Patient was admitted to non-VA hospital for A-fib. Treated with Amiodarone drip and cardioversion.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=5) | Intervention Group (N=5)
Not Fasted (General disorders) | 0 (0) | 1 (1) — Patient was not fasted at baseline visit. Patient completed fast blood draw on first day of intervention instead of during baseline visit. He confirmed he was fasted.

LIMITATIONS AND CAVEATS:
Participation in this study hinged on recruitment into the parent study which was delayed due to various location and staff changes and early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-07-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT02275819/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT02275819/Prot_SAP_001.pdf